CLINICAL TRIAL: NCT00631033
Title: Diazoxide-mediated Insulin Suppression in Hyperinsulinemic Obese Men, Part III
Brief Title: DZX Mediated Insulin Suppression in Obese Men
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LTC-511-230108
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Obesity
Keywords: obesity; hyperinsulinism; diazoxide; metformin
MeSH Terms: conditions — Obesity; Hyperinsulinism | interventions — Diazoxide; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 2 (Experimental): Diazoxide
  Interventions: Drug: Diazoxide
- 3 (Experimental): Metformin + Diazoxide
  Interventions: Drug: Metformin + Diazoxide

INTERVENTIONS:
Drug: Placebo
  Arms: 1
Drug: Diazoxide
  Arms: 2
Drug: Metformin + Diazoxide
  Arms: 3

SUMMARY:
The purpose of this study is to determine whether there is an additive effect of metformine on the weight reduction of obese hyperinsulinemic men who are treated with diazoxide.

ELIGIBILITY:
Inclusion Criteria:

* male
* age 25-50 years
* BMI 30-35 kg/m2
* stable body weight during 3 months before the start of the study
* glucose <= 6.0 mmol/L
* C-peptide >= 1.0 nmol/L
* HbA1c <= 6.0%

Exclusion Criteria:

* comorbidity
* medication
* serum creatinine > 120 micromol/L
* liver enzymes > 2 times upper limits of normal
* gout
* alcohol use > 2 alcoholic drinks a day
* drug abuse
* cessation of smoking less than 6 months ago

Ages: 25 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2008-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rijnstate Hospital, Arnhem, Netherlands

REFERENCES:
- [Derived] Loves S, van Groningen L, Filius M, Mekking M, Brandon T, Tack CJ, Hermus A, de Boer H. High-Dose, Diazoxide-Mediated Insulin Suppression Boosts Weight Loss Induced by Lifestyle Intervention. J Clin Endocrinol Metab. 2018 Nov 1;103(11):4014-4022. doi: 10.1210/jc.2018-01147. PMID 30202851
- [Derived] Loves S, van Groningen L, Filius M, Mekking M, Brandon T, Tack CJ, Hermus A, de Boer H. Effects of Diazoxide-Mediated Insulin Suppression on Glucose and Lipid Metabolism in Nondiabetic Obese Men. J Clin Endocrinol Metab. 2018 Jun 1;103(6):2346-2353. doi: 10.1210/jc.2018-00161. PMID 29618011